CLINICAL TRIAL: NCT02220946
Title: Effect of Vaginal Electrical Stimulation on Female Sexual Dysfunction
Acronym: EVESOFS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, serdar aydin, MD, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EVESFDS
Record Dates: First submitted 2014-08-17; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Female Sexual Dysfunction
Keywords: Vaginal Electrical Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaginal Electrical Stimulation (Active Comparator): A vaginal probe inserted, and a medium frequency (50 Hz) alternating current was administered for 5 seconds on, 5 seconds off the intensity of the current was started at 0 mA, and gradually increased until pelvic muscle contractions was observed, then increased according to patient tolerance. Each patient received a 20 minute session once a week for total 8 sessions
  Interventions: Device: Vaginal Electrical Stimulation
- plasebo (Placebo Comparator): sham electrical stimulation

INTERVENTIONS:
Device: Vaginal Electrical Stimulation — A vaginal probe inserted, and a medium frequency (50 Hz) alternating current was administered for 5 seconds on, 5 seconds off. the intensity of the current was started at 0 mA, and gradually increased until pelvic muscle contractions was observed, then increased according to patient tolerance. each patient received a 20 minute session once a week for total 8 session
  Other Names: MyoBravo Electrical Stimulation Device
  Arms: Vaginal Electrical Stimulation

SUMMARY:
vaginal electrical stimulation improves female sexual dysfunction

ELIGIBILITY:
Inclusion Criteria:

* women with complaint of sexual dysfunction at any part of sexual cycle

Exclusion Criteria:

* pregnancy previous gynecologic surgery pelvic organ prolapsus greater than stage 1 women with neurological disease and anatomical defect women with anatomical defect

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in on domains and total score of Female Sexual Function Index (FSFI) at week 8 | Baseline, Week 8

SECONDARY OUTCOMES:
Change from baseline in power, endurance, dynamic endurance and fast contractions on the PERFECT scheme at week 8 | Baseline, Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetric and Gynecology, Bezmialem Vakif University, Istanbul, Turkey (Türkiye)